CLINICAL TRIAL: NCT02767791
Title: Auriculotherapy and Acupuncture's Treatment for Chemotherapy-induced Nausea and Vomiting (CINV)
Acronym: NVCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/34; 2015-A01988-41 (Other: ANSM)
Record Dates: First submitted 2016-05-04; First posted 2016-05-10 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Acupuncture Therapy; Auriculotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Acupuncture (Active Comparator): Acupuncture wrist 6
  Interventions: Other: Acupuncture
- Auriculotherapy (Active Comparator): Auriculotherapy
  Interventions: Other: Auriculotherapy
- Auriculotherapy and acupuncture (Experimental): Auriculotherapy and acupuncture
  Interventions: Other: Acupuncture; Other: Auriculotherapy
- No treatment (No Intervention): No treatment

INTERVENTIONS:
Other: Acupuncture — Acupuncture
  Arms: Acupuncture; Auriculotherapy and acupuncture
Other: Auriculotherapy — Auriculotherapy
  Arms: Auriculotherapy; Auriculotherapy and acupuncture

SUMMARY:
The management of chemotherapy-induced nausea and vomiting (CINV) has evolved in recent years and became less frequent. CINV include early (occurring within 24 hours of chemotherapy administration) and delayed (occurring within 4 days after chemotherapy) nausea and vomiting.

Preventive treatment, such as Glucocorticoids, 5-hydroxytryptamine type 3 (5-HT3) receptor antagonists and neurokinin 1 (NK1) receptor antagonists, are administered according to the classification in 4 grades of expected CINV

* Very low: <10% occurrence of CINV;
* Low: 10 to 30% occurrence of CINV;
* Average: 30 to 90% occurrence of CINV;
* High: > 90% occurrence of CINV. These treatments have been the subject of recommendations. Despite these available treatments, some patients still complain of vomiting, or more frequently nausea and loss of appetite.

Meanwhile, Chinese acupuncture has proven effective on the prevention of CINV as complementary treatment, mainly in the acute phase and to a lesser extent in the delayed phase. The most common points are Pericardium 6 (wrist) treated with conventional acupuncture needles, electro-acupuncture or acupressure.

Auriculotherapy (ear acupuncture) has proven effective on nausea of pregnancy and postoperative nausea, but, to our knowledge, there are no studies published on the effect of auriculotherapy on CINV.

These complementary treatments have virtually no side effects. In our institution, a simple treatment of acupuncture (2 points Pericardium 6 treated) and auriculotherapy (2 auricular point treated) is regularly use in patients who present CINV despite preventive treatment and most of them are relieved.

The investigators propose a clinical trial in this population to assess symptoms improvement in patients presenting CINV after their first administration of chemotherapy despite adapted preventive treatment. Experimental treatment with semi-permanent needles takes place during administration of the second session of chemotherapy. CINV are evaluated through the (MAT) score that measures the frequency and intensity of nausea and vomiting in the 24 hours following the session and during the 4 days after administration Chemotherapy.

Multinational Association of Supportive Care in Cancer Antiemesis Tool (MASCC), Http://www.MASCC.org/.

ELIGIBILITY:
Inclusion Criteria:

* out-patient chemotherapy
* treated nausea vomiting induced by chemotherapy (NVIC)

Exclusion Criteria:

* prior treatment with acupuncture and or auriculotherapy for NVIC
* no conventional treatment for NVIC like phytotherapy and homeopathy
* radiotherapy (five days before and 5 days after chemotherapy)
* MRI in the five days after first visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Digital Scale for nausea | 1 day
  Digital Scale for nausea (H24 MAT score)

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Michel-Cherqui, MD, Principal Investigator — Hopital Foch
Locations (5):
- France (5):
  - Centre hospitalier de Gonesse, Gonesse
  - René Huguenin, Saint-Cloud
  - Centre spécilaisé en cancérologie Paris Nord, Sarcelles
  - Clinique de l'Estrée, Stains
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michel-Cherqui M, Ma S, Bacrie J, Huguet S, Lemaire N, Le Guen M, Fischler M. Auriculotherapy and acupuncture treatments for chemotherapy-induced nausea and vomiting: a multicenter clinical trial. Support Care Cancer. 2024 Jul 31;32(8):560. doi: 10.1007/s00520-024-08768-w. PMID 39085664